CLINICAL TRIAL: NCT03253770
Title: Use of a Hand-held Digital Cognitive Aid in Simulated Cardiac Arrest.
Acronym: SIMMAX2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, CEJKA Jean-Christophe, MD, PhD, MEng, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIMMAX2
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Cardiac Arrest
Keywords: Cognitive Aid
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital Cognitive Aid (Experimental): The digital cognitive aid is designed as a smartphone app. Intervention : cognitive aid in the hand of the leader during crises management.
  Interventions: Device: SIMMAX2
- No digital aid (Experimental): No cognitive aid in the hand of the leader during crises management. Intervention : no cognitive aid in the hand of the leader during crises management.
  Interventions: Device: SIMMAX2
- Paper Cognitive Aid (Experimental): The paper cognitive aid is the document officially recommended to be used in case of crises by the French Society of Anaesthesia and Intensive Care.
  Intervention : paper cognitive aid in the hand of the leader during crises management.
  Interventions: Device: SIMMAX2

INTERVENTIONS:
Device: SIMMAX2 — Digital cognitive aid or paper cognitive aid during the management of a cardiac arrest in the recovery room or in the delivery room.

SUMMARY:
Cardiac arrest is one of the most stressful situations to be managed. Our first study (MAX, accepted for publication BJA) clearly showed that it could not be compared to other urgent and stressful situations (malignant hyperthermia, anaphylactic shock, acute toxicity of local anesthetics, severe and symptomatic hyperkaliemia) whose management was significantly improved with the help of a digital cognitive aid.

The present study exclusively deals with the management of cardiac arrest (recovery ward, or in the delivery room.) with the second generation of our digital cognitive aid, and explores new insights on how to better manage cardiac arrest with a digital cognitive aid in the hand of the leader.

DETAILED DESCRIPTION:
" Errare humanum est ", to err is human. This Latin saying attributed to Seneca shows that since the dawn of time, human beings are aware that managing complex situations will always be an inexhaustible source of mistakes. This is particularly true in anesthesia and intensive care in which situations are often complex and stressful, thus leading to mistakes or inadequate management. Improvement might arise from the use of cognitive aids.

In a first study (MAX, accepted for publication BJA) the investigators designed a smartphone application including 5 scenarios of anesthesia and intensive care crises (malignant hyperthermia, anaphylactic shock, acute toxicity of local anesthetics, severe and symptomatic hyperkaliemia, ventricular fibrillation), designed to be used in the hand of the leader managing the crises. Technical and non technical skills were improved in 4 out of 5 scenarios. Cardiac arrest (ventricular fibrillation) clearly happened to be a different situation compared to other crises, and no improvement could be measured with our cognitive aid.

The present study exclusively deals with the management of cardiac arrest (man in recovery ward, pregnant woman in the delivery room) with the second generation of our digital cognitive aid, and explores new insights on how to better manage cardiac arrest with a digital cognitive aid in the hand of the leader.

ELIGIBILITY:
Inclusion Criteria:•

* Resident Physicians training in Anesthesia/Intensive care (same specialization in France), year 1 to 5 (out of 5)
* to be familiar with our simulation centre (at least passed once as a resident)

Exclusion Criteria:

* no experience in simulation training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Technical Performance as compared to a Reference Task List | [ Time Frame: Time 0-30 min ]
  Number of tasks successfully performed, rated on remote video review

SECONDARY OUTCOMES:
Non technical skills performance | [ Time Frame: Time 0-30 min ]
  As measured by the Ottawa score, rated on remote video review

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Lyonnais d'Enseignement par la Simulation en Santé, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided